CLINICAL TRIAL: NCT02300259
Title: A Study to Determine the Effect of CYP3A Inhibition on the Pharmacokinetics of LY2623091 and the Effect of LY2623091 on the Pharmacokinetics of CYP3A Substrates in Healthy Subjects
Brief Title: A Study of LY2623091 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15523; I7T-MC-RMAG (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-11-20; First posted 2014-11-24 (Estimated); Results first posted 2020-06-26 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Itraconazole; Simvastatin; Tadalafil; Diltiazem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- LY2623091 (Group 1) (Experimental): LY2623091 administered orally once on Day 1 of Period 1.
  Interventions: Drug: LY2623091
- Itraconazole + LY2623091 (Group 1) (Experimental): 200 mg itraconazole administered orally twice daily on Day 1 of Period 2 and once daily on Days 2 - 20 of Period 2. Single oral dose of LY2623091 coadministered on Day 6 of Period 2.
  Interventions: Drug: LY2623091; Drug: Itraconazole
- Simvastatin (Group 2) (Experimental): 20 mg simvastatin administered orally once daily on Day 1.
  Interventions: Drug: Simvastatin
- LY2623091 + Simvastatin (Group 2) (Experimental): LY2623091 administered orally once daily on Days 3 - 13. Single oral dose of 20 mg simvastatin coadministered on Day 12.
  Interventions: Drug: LY2623091; Drug: Simvastatin
- Tadalafil (Group 3) (Experimental): 5 mg tadalafil administered on Day 1 of Period 1. Arm is contingent on interim results from Groups 1 and 2.
  Interventions: Drug: Tadalafil
- Tadalafil + LY2623091 (Group 3) (Experimental): LY2623091 administered orally once daily on Day 1 up to Day 15 of Period 2. 5 mg tadalafil co-administered once daily on Day 10 of Period 2. Arm is contingent on interim results from Groups 1 and 2.
  Interventions: Drug: LY2623091; Drug: Tadalafil
- LY2623091 (Group 4) (Experimental): LY2623091 administered orally once on Day 1 of Period 1. Arm is contingent on interim results from Groups 1 and 2.
  Interventions: Drug: LY2623091
- Diltiazem + LY2623091 (Group 4) (Experimental): 240 mg diltiazem administered once daily on Days 1 to 13 of Period 2. Single oral dose of LY2623091 coadministered on Day 4 of Period 2. Arm is contingent on interim results from Groups 1 and 2.
  Interventions: Drug: LY2623091; Drug: Diltiazem

INTERVENTIONS:
Drug: LY2623091 — Administered orally
  Arms: Diltiazem + LY2623091 (Group 4); Itraconazole + LY2623091 (Group 1); LY2623091 (Group 1); LY2623091 (Group 4); LY2623091 + Simvastatin (Group 2); Tadalafil + LY2623091 (Group 3)
Drug: Itraconazole — Administered orally
  Arms: Itraconazole + LY2623091 (Group 1)
Drug: Simvastatin — Administered orally
  Arms: LY2623091 + Simvastatin (Group 2); Simvastatin (Group 2)
Drug: Tadalafil — Administered orally
  Arms: Tadalafil (Group 3); Tadalafil + LY2623091 (Group 3)
Drug: Diltiazem — Administered orally
  Arms: Diltiazem + LY2623091 (Group 4)

SUMMARY:
The first purpose of this study is to evaluate the effect of itraconazole (and possibly diltiazem) on the amount of LY2623091 in the blood stream and how long the body takes to get rid of it.

The second purpose of the study is to evaluate the effect of LY2623091 on the amount of simvastatin (and possibly tadalafil) in the blood stream and how long the body takes to get rid of it.

The safety and tolerability of LY2623091 when given with itraconazole, simvastatin and diltiazem or tadalafil will be evaluated.

There will be three groups of participants in this study. Results from Groups 1 and 2 will be analyzed during the study to determine whether to enroll participants in Group 3 or 4. The study is expected to last up to 40 days from the first dose to follow-up (inclusive). Screening may occur up to 28 days prior to enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants as determined by medical history, physical examination, clinical laboratory tests, and electrocardiograms (ECGs).
* Have a body mass index (BMI) between 18 and 32.0 kilograms per square meter (kg/m^2) inclusive, at screening
* Female participants must be of non-childbearing potential

Exclusion Criteria:

* In the opinion of the investigator or sponsor, are unsuitable for inclusion in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Inc, Daytona Beach, Florida, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study planned to enroll 3 groups. After Groups 1 and 2 were enrolled, data from Group 2 were analyzed according to a pre-specified algorithm. Results met criteria to enroll Group 4. (Group 3 was not enrolled.)
Groups:
- LY2623091 + Itraconazole (Group 1): Period 1: Single oral dose of 6 mg LY2623091 on Day 1.
  Period 2: Oral doses of 200 mg itraconazole twice daily (BID) on Day 1 and then once daily (QD) on Days 2 to 20 with a single oral dose of 6 mg LY2623091 coadministered on Day 6.
- Simvastatin + LY2623091 (Group 2): Single oral dose of 20 mg simvastatin on Day 1 followed by oral doses of 24.5 mg LY2623091 QD on Days 3 to 13, with a single oral dose of 20 mg simvastatin coadministered on Day 12.
- LY2623091 + Diltiazem (Group 4): Period 1: Single oral dose of 6 mg LY2623091 on Day 1.
  Period 2: Oral doses of 240 mg diltiazem extended release QD on Days 1 to 13, with a single oral dose of 6 mg LY2623091 coadministered on Day 4.
Period: Period 1
Arm/Group | LY2623091 + Itraconazole (Group 1) | Simvastatin + LY2623091 (Group 2) | LY2623091 + Diltiazem (Group 4)
Started | 16 | 16 | 16
Received at Least One Dose of Study Drug | 16 | 16 | 16
Completed | 16 | 16 | 14
Not Completed | 0 | 0 | 2
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1
Period: Period 2
Arm/Group | LY2623091 + Itraconazole (Group 1) | Simvastatin + LY2623091 (Group 2) | LY2623091 + Diltiazem (Group 4)
Started | 16 | 0 (There was no period 2 for Group 2.) | 14
Completed | 15 | 0 | 13
Not Completed | 1 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- LY2623091 + Itraconazole (Group 1): Period 1: Single oral dose of 6 mg LY2623091 on Day 1.
  Period 2: Oral doses of 200 mg itraconazole BID on Day 1 and then QD on Days 2 to 20 with a single oral dose of 6 mg LY2623091 coadministered on Day 6.
- Total: Total of all reporting groups
Arm/Group | LY2623091 + Itraconazole (Group 1) | Simvastatin + LY2623091 (Group 2) | LY2623091 + Diltiazem (Group 4) | Total
Number analyzed (Participants) | 16 | 16 | 16 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (9.4) | 37.8 (10.1) | 39.2 (9.3) | 39.7 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 7 | 13
  Male | 12 | 14 | 9 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 8 | 8 | 25
  Not Hispanic or Latino | 7 | 8 | 8 | 23
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 5 | 6 | 16
  White | 10 | 9 | 10 | 29
  More than one race | 1 | 2 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 16 | 48

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics: Maximum Drug Concentration (Cmax) of LY2623091
Time Frame: Group 1 (Days 1 and 6) Group 4 (Days 1 and 4): Predose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 96, 120, 144, 168, 192, 216, 240 hours (hr) postdose; additionally for Group 1 (Day 6): 264, 288, 312, 336, 360 hr postdose
Population: All participants in Groups 1 and 4 who received at least one dose of study drug and had evaluable Cmax results.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Groups:
- LY2623091 (Group 1): Period 1: Single oral dose of 6 mg LY2623091 on Day 1.
- Itraconazole + LY2623091 (Group 1): Period 2: Oral doses of 200 mg itraconazole BID on Day 1 and then QD on Days 2 to 20 with a single oral dose of 6 mg LY2623091 coadministered on Day 6.
- LY2623091 (Group 4): Period 1: Single oral dose of 6 mg LY2623091 on Day 1.
  .
- Diltiazem + LY2623091 (Group 4): Period 2: Oral doses of 240 mg diltiazem extended release QD on Days 1 to 13, with a single oral dose of 6 mg LY2623091 coadministered on Day 4.
Arm/Group | LY2623091 (Group 1) | Itraconazole + LY2623091 (Group 1) | LY2623091 (Group 4) | Diltiazem + LY2623091 (Group 4)
Number analyzed (Participants) | 16 | 16 | 16 | 14
nanograms per milliliter (ng/mL) | 61.9 (21) | 66.9 (27) | 61.8 (34) | 64.2 (30)

2. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-infinity]) of LY2623091
Time Frame: as for outcome 1
Population: All participants in Groups 1 and 4 who received at least one dose of study drug and had evaluable AUC(0-infinity) results.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour/milliliter (ng*h/mL)
Groups:
- LY2623091 (Group 4): Period 1: Single oral dose of 6 mg LY2623091 on Day 1.
Arm/Group | LY2623091 (Group 1) | Itraconazole + LY2623091 (Group 1) | LY2623091 (Group 4) | Diltiazem + LY2623091 (Group 4)
Number analyzed (Participants) | 16 | 16 | 16 | 14
nanograms*hour/milliliter (ng*h/mL) | 2540 (27) | 5660 (31) | 2390 (39) | 3360 (43)

3. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Time Zero to Time T, Where T is the Last Time Point With a Measurable Concentration (AUC[0-tlast]) of LY2623091
Time Frame: as for outcome 1
Population: All participants in Groups 1 and 4 who received at least one dose of study drug and had evaluable AUC(0-tlast) results.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | LY2623091 (Group 1) | Itraconazole + LY2623091 (Group 1) | LY2623091 (Group 4) | Diltiazem + LY2623091 (Group 4)
Number analyzed (Participants) | 16 | 15 | 16 | 14
ng*hr/mL | 2480 (27) | 5240 (31) | 2340 (39) | 3130 (40)

4. Primary Outcome: Pharmacokinetics: Maximum Drug Concentration (Cmax) of Simvastatin and Simvastatin Acid
Time Frame: Days 1 and 12: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12 hours postdose
Population: All participants in Group 2 who received at least one dose of study drug and had evaluable Cmax results.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Simvastatin (Group 2): Single oral dose of 20 mg simvastatin on Day 1.
- LY2623091 + Simvastatin (Group 2): Oral doses of 24.5 mg LY2623091 QD on Days 3 to 13, with a single oral dose of 20 mg simvastatin coadministered on Day 12.
Arm/Group | Simvastatin (Group 2) | LY2623091 + Simvastatin (Group 2)
Number analyzed (Participants) | 16 | 16
ng/mL
  Simvastatin | 7.78 (63) | 9.89 (45)
  Simvastatin Acid | 0.720 (41) | 0.877 (55)

5. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Zero to Infinity (AUC[0-infinity]) of Simvastatin and Simvastatin Acid
Time Frame: Days 1 and 12: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12 hours postdose
Population: All participants in Group 2 who received at least one dose of study drug and had evaluable AUC(0-infinity) results.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Groups:
- LY2623091 + Simvastatin: Oral doses of 24.5 mg LY2623091 QD on Days 3 to 13, with a single oral dose of 20 mg simvastatin coadministered on Day 12.
Arm/Group | Simvastatin (Group 2) | LY2623091 + Simvastatin
Number analyzed (Participants) | 16 | 16
ng*h/mL
  Simvastatin | 17.4 (48) | 24.1 (34)
  Simvastatin Acid: number analyzed (Participants) | 11 | 10
  Simvastatin Acid | 7.15 (56) | 8.88 (77)

6. Primary Outcome: Pharmacokinetics: Area Under the Concentration Versus Time Curve From Time Zero to Time T, Where T is the Last Time Point With a Measurable Concentration (AUC[0-tlast]) of Simvastatin and Simvastatin Acid
Time Frame: Days 1 and 12: Predose, 0.5, 1, 2, 3, 4, 6, 8, 12 hours postdose
Population: All participants in Group 2 who received at least one dose of study drug and had evaluable AUC(0-tlast) results.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Simvastatin (Group 2) | LY2623091 + Simvastatin
Number analyzed (Participants) | 16 | 16
ng*hr/mL
  Simvastatin | 16.5 (49) | 23.0 (34)
  Simvastatin Acid | 5.42 (48) | 6.87 (87)

ADVERSE EVENTS:
Description: Includes serious adverse events (SAEs) and all other non-serious adverse events (AEs) that met the frequency threshold regardless of causality.
Groups:
- Itraconazole (Group 1): Period 2: Oral doses of 200 mg itraconazole BID on Days 1 through 5.
- Itraconazole + LY2623091 (Group 1): Period 2: Oral doses of 200 mg itraconazole and 6 mg LY2623091 coadministered once on Day 6.
- LY2623091 (Group 2): Oral doses of 24.5 mg LY2623091 QD on Days 3 to 11.
- LY2623091 + Simvastatin (Group 2): Oral doses of 24.5 mg LY2623091 and 20 mg simvastatin coadministered once on Day 12.
- Diltiazem (Group 4): Period 2: Oral doses of 240 mg diltiazem extended release QD on Days 1 through 3.
- Diltiazem + LY2623091 (Group 4): Period 2: Oral doses of 240 mg diltiazem extended release and 6 mg LY2623091 coadministered once on Day 4.
Arm/Group | LY2623091 (Group 1) | Itraconazole (Group 1) | Itraconazole + LY2623091 (Group 1) | Simvastatin (Group 2) | LY2623091 (Group 2) | LY2623091 + Simvastatin (Group 2) | LY2623091 (Group 4) | Diltiazem (Group 4) | Diltiazem + LY2623091 (Group 4)
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/16 | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 0/16 | 3/16 | 6/16 | 0/16 | 4/16 | 1/16 | 3/16 | 1/14 | 1/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LY2623091 (Group 1) (N=16) | Itraconazole (Group 1) (N=16) | Itraconazole + LY2623091 (Group 1) (N=16) | Simvastatin (Group 2) (N=16) | LY2623091 (Group 2) (N=16) | LY2623091 + Simvastatin (Group 2) (N=16) | LY2623091 (Group 4) (N=16) | Diltiazem (Group 4) (N=14) | Diltiazem + LY2623091 (Group 4) (N=14)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cyst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days